CLINICAL TRIAL: NCT05711602
Title: Influence of the Pilates Method on the Physical and Mental Health of People With Type II Diabetes Mellitus.
Brief Title: The Physical and Mental Health of People With Type II Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Physiotherapy, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University_of_Jaén
Record Dates: First submitted 2023-01-21; First posted 2023-02-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Adult ALL; Diabete Type 2
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Diabetes Mellitus, Type 2 | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to the groups will be of simple random type and hidden. Those responsible for admitting patients to the intervention phase will not know what group has been assigned each. This assignment will be made in advance by a researcher who will not intervene in the later stages of evaluation, intervention, data recording and elaboration of database. The assignment will be communicated through sealed and totally opaque envelopes.
  All measurements given above will be made both to the control group and to the experimental group just prior to the start of the intervention, and immediately after and six months after the end of this period, and the results will be recorded in a data record
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental): This group receives physical training based on pilates exercises
  Interventions: Other: Pilates
- No intervention group (No Intervention): This group does not receive any treatment

INTERVENTIONS:
Other: Pilates — raining based on a basic level Pilates exercise program will be as follows: A duration of weeks with a frequency of 2 sessions a week and with a duration of 55 minutes each. The exercises to be performed will be divided into three distinct phases: warm-up, lasting 15 minutes; Main part with a duration of 30 minutes and the return to calm, based mostly on stretching and with a duration of 10 minutes. The repetitions of the exercises will be between 5 and 10 according to the difficulty.
  Arms: Pilates group

SUMMARY:
To analyze the effects of a Pilates exercise program on physical and mental health in people with type II diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 2 arms (Control group and experimental group), in which a pre-treatment-postest design has been used.

The study will define two groups:

* A control group (CG) that will not be submitted to treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity and will be given a guide to recommendations for promoting physical activity.
* An experimental group (GE) that after an initial evaluation will undergo a physical training program based on Pilates exercises.

Once the intervention is finished, it will be submitted to a final evaluation to see if there is a difference or not with the results obtained at the beginning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Not participating in an exercise program
* That they were able to carry out the different selected questionnaires.

Exclusion Criteria:

* Contraindications for performing physical tests
* Illnesses that limit static and dynamic balance and physical activity
* Central or peripheral vestibular or nervous disorders.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Dynamometer | Up to twelve weeks
  Dynamometer will be employed to assess hand grip stregth.
Blood Glucose Concentration | Up to twelve weeks
  Capillary blood glucose monitoring is the primary tool for monitoring blood glucose levels at any time of day. It involves a small fingertip prick to check blood sugar levels at a specific time of day. This procedure requires a pen containing a fine needle or lancet, test strips, and a glucose meter (glucometer). Reference values vary depending on the time of sample collection: preprandial 80-130 mg/dL and postprandial <180 mg/dL. In Spain, this measurement is performed among older adults with type 2 diabetes mellitus.
BMI (Body Mass Index) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
TUG (Timed Up and Go test) | Up to twelve weeks
  Is a simple test used to assess a person's mobility and physical function
Chair sit and reach test | Up to twelve weeks
  To test low back and hamstring flexibility.
Back scratch test | Up to twelve weeks
  To measure general shoulder range of motion.
Height | Up to twelve weeks
  The distance between the lowest and highest points of a person standing upright.
BBS (the Berg Balance Scale) | Up to twelve weeks
  Used to measure balance

CONTACTS AND LOCATIONS:
Locations (1):
- U.E.D. Virgen de la Capilla, Jaén, Spain